CLINICAL TRIAL: NCT01638052
Title: Great Auricular Nerve Block for Children Undergoing Tympanomastoid Surgery: Does the Addition of Clonidine Increase the Duration of Postoperative Analgesia?
Brief Title: Great Auricular Nerve Block for Children Undergoing Tympanomastoid Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CMH IRB 2005-12645
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2012-07

CONDITIONS: Tympanomastoid Surgery; Cochlear Implant; Mastoidectomy; Cholesteatoma
Keywords: Tympanomastoid Surgery; Cochlear Implant; Mastoidectomy; Cholesteatoma; Pediatrics; Clonidine; Bupivacaine; Greater Auricular Nerve Block; Regional Anesthesia
MeSH Terms: conditions — Cholesteatoma | interventions — Bupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.25% Bupivacaine (No Intervention): This is our standard of care concentration
- 0.25% Bupivacaine + Clonidine (Experimental): These are not two separate drugs, but a mixture of Bupivacaine and Clonidine.
  Interventions: Drug: 0.25% Bupivacaine + Clonidine

INTERVENTIONS:
Drug: 0.25% Bupivacaine + Clonidine — Patients will receive 2mL of 0.25% bupivacaine with 2mcg/ml of clonidine
  Other Names: Marcaine
  Arms: 0.25% Bupivacaine + Clonidine

SUMMARY:
The investigators goal is to determine the efficacy and duration of analgesia with the addition of Clonidine, an alpha-2 agonist, to local anesthetic blockade using bupivacaine, of the great auricular nerve in children undergoing tympanomastoid surgery.

DETAILED DESCRIPTION:
The surgical anesthesia during the operative procedure will be maintained using volatile anesthetics. No prophylactic dexamethasone or ondansetron would be provided to any patients in either group. Anesthesia will be discontinued at the end of the procedure and the patient will be extubated once standard extubation criteria have been met. Patients will be then taken to the postoperative recovery room where they will be evaluated for pain and discomfort by a blinded observer using the CHIPPS (Children and Infants Postoperative Pain Scale). If two consecutive pain scores at 5 minute intervals is >6, they will be rescued with incremental doses of 0.05 mg/kg of intravenous morphine required to reach a score of <6. The number of rescue doses as well as the pain scores will be documented. These patients will be also observed for the presence of nausea/vomiting. Any patient who vomits more than two times will be rescued with ondansetron 0.1 mg/kg intravenously. All patients will be continued to be evaluated in the 23 hour unit. Pain and side effects will be assessed for the next 6 hours or until discharge from the 23 hour observation facility. Standard doses of acetaminophen with codeine will be provided for pain relief in the 23 hour observational unit, as well as on discharge. The number of doses of acetaminophen with codeine will be recorded. Time to discharge from the hospital will also be noted. A questionnaire designed to address parent/patient satisfaction will be utilized and will allude to the need for rescue analgesia and the need for any other additional analgesics provided. The use of any additional rescue pain medication will be provided to the families at the time of discharge. A follow-up phone call will be made in 24 hours to note the information provided on the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age 1-18 years
* tympanomastoid surgery (cochlear implant, mastoidectomy, cholesteatoma surgery)
* ASA I, II
* informed consent and assent obtained

Exclusion Criteria:

* allergic to local anesthestic
* taking chronic aspirin or Ibuprofen therapy
* ASA IV
* history of clinically important renal, hepatic, respiratory, cardiac, or neurological conditions
* Patients who have cardiovascular surgery other than an atrial septal defect or a ventricular septal defect, or who have undergone complete corrective intracardiac repair of congenital heart disease.
* Informed consent not obtained
* Patients expected to receive dexamethasone or ondansetron intra-operative

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santhanam Suresh, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Suresh S, Barcelona SL, Young NM, Seligman I, Heffner CL, Cote CJ. Postoperative pain relief in children undergoing tympanomastoid surgery: is a regional block better than opioids? Anesth Analg. 2002 Apr;94(4):859-62, table of contents. doi: 10.1097/00000539-200204000-00015. PMID 11916785
- [Background] Wheeler M, Patel A, Suresh S, Roth AG, Birmingham PK, Heffner CL, Cote CJ. The addition of clonidine 2 microg.kg-1 does not enhance the postoperative analgesia of a caudal block using 0.125% bupivacaine and epinephrine 1:200,000 in children: a prospective, double-blind, randomized study. Paediatr Anaesth. 2005 Jun;15(6):476-83. doi: 10.1111/j.1460-9592.2005.01481.x. PMID 15910348

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.25% Bupivacaine + Clonidine: These are not two separate drugs, but a mixture of Bupivacaine and Clonidine.
  0.25% Bupivacaine + Clonidine : Patients will receive 2mL of 0.25% bupivacaine with 2mcg/ml of clonidine
Period: Overall Study
Arm/Group | 0.25% Bupivacaine | 0.25% Bupivacaine + Clonidine
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.25% Bupivacaine | 0.25% Bupivacaine + Clonidine | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Full Range); unit: years] | 6.9 [1 to 17] | 7.5 [1 to 18] | 7.2 [1 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Average Observer-Rated Patient Pain Scores
Description: Patients will be observed with behaviors rated at regular time intervals using the CHIPPS (Children and Infants Postoperative Pain Scale) pain survey. The CHIPPS scale values range from a minimum of 0 (no pain, better outcome) to a maximum of 10 (worst pain, worse outcome).
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.25% Bupivacaine | 0.25% Bupivacaine + Clonidine
Number analyzed (Participants) | 28 | 28
units on a scale | 2 (1.05) | 1.9 (1.05)

2. Secondary Outcome: Number of Participants With Nausea/Vomiting
Description: Incidence of nausea/vomiting during 24 hour observation
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Bupivacaine | 0.25% Bupivacaine + Clonidine
Number analyzed (Participants) | 28 | 28
Participants | 14 | 10

3. Secondary Outcome: Number of Participants Requiring Use of Rescue Analgesic Medication in the Initial 24 Hours Postoperatively
Description: Count of participants who will require use of rescue analgesic medication in the initial 24 hours postoperatively as recorded in the hospital or by parents at home following discharge.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% Bupivacaine | 0.25% Bupivacaine + Clonidine
Number analyzed (Participants) | 28 | 28
Participants | 18 | 22

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | 0.25% Bupivacaine | 0.25% Bupivacaine + Clonidine
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes